CLINICAL TRIAL: NCT02541916
Title: Liver Immune Tolerance Marker Utilization Study
Acronym: LITMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Gary A Levy, O. Ont. MD. FRCP AGAF, Principle Investigator, Professor, O. Ont. MD. FRCP AGAF, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Tol002
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Immunosuppression; Immune Tolerance
Keywords: Transplantation Tolerance; Immune Tolerance; Transplantation; Liver Transplantation; Biological Markers; Gene Expression; Immunosuppression; Immunology; Multiplex Polymerase Chain Reaction; Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Controlled weaning of immunosuppression (Experimental): Participants who are found to have the tolerance gene expression profile during phase 1 of the study will undergo closely monitored immunosuppression weaning during phase 2.
  Interventions: Other: Controlled weaning of immunosuppression

INTERVENTIONS:
Other: Controlled weaning of immunosuppression — At week 0 patients have liver biopsy and liver functional tests (LFTs). Week 1-4 medication reduction to 1.5mg Tacrolimus (Tac) daily or 150mg Cyclosporine A (CsA). At week 4 LFTs. Week 5-8 medication reduction to 1mg Tac / 100mg CsA. Week 8 LFTs. Week 9-12 reduction to 0.5mg Tac/ 50mg CsA. Week 12 LFTs. Week 13-16 reduction to 0mg. Week 16 liver biopsy & LFTs. Weekly LFTs performed Week 17-20. Monthly LFTs for the next 3 months. LFTs every 3 months for monitoring.

SUMMARY:
The purpose of this study is to validate and test a tolerance gene expression profile for the identification of operationally tolerant liver transplant recipients, allowing for the successful withdrawal of immunosuppression without rejection in these patients.

DETAILED DESCRIPTION:
Previous pre-clinical work in the Levy Lab identified a novel biomarker gene set for the identification of tolerance in murine models of rapamycin-induced cardiac tolerance and spontaneous hepatic tolerance. Validation of this gene expression tolerance biomarker in operationally tolerant patients is now required for its implementation in the clinical setting. This proposal intends to validate and test our pre-clinically established tolerance gene expression biomarker in the clinical setting in order to translate our findings into improving the length and quality of life of transplant patients in the clinic.

The investigators hypothesize that a distinct gene expression profile expressed in the peripheral blood will identify operationally tolerant liver transplant recipients, allowing for the successful withdrawal of immunosuppression in these patients. Our study aims are: (I) To validate the pre-clinical gene expression profile for the identification of operationally tolerant liver recipients in plasma peripheral blood mononuclear cells (PBMCs) (2) To determine that the gene expression profile in the PBMCs is the same as the intra-graft gene expression profile (3) To demonstrate that liver transplant recipients with the tolerant gene expression profile can be safely weaned off of immunosuppression.

This proof of principle study will be conducted in two phases at the Toronto General Hospital (TGH) Phase 1 will address study aims 1 and 2, and phase 2 will address study aim 3. Potential participants will be screened and selected following predefined eligibility criteria. Eligible participants will undergo an informed consent process. The primary goal of this study is to validate the pre-clinical tolerant gene expression profile that will allow for the identification of tolerant liver recipients and for the monitored weaning off immunosuppression in these tolerant patients.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, patients must:

  1. Be between 18 and 65 years of age.
  2. Be recipients of a hepatic allograft.
  3. Be less than 3 months post-transplant and be experiencing rejection, or be a minimum of 3 months post-transplant with or without presently experiencing rejection.
  4. Be healthy live liver donors

Exclusion Criteria:

* Patients with the following conditions may not participate in the study:

  1. Patients under the age of 18 and over the age of 65.
  2. Patients who are positive for Human Immunodeficiency Virus (HIV),
  3. Patients who have detectable levels of HCV RNA, and HBV DNA, at the time of enrollment.
  4. Patients who have a combined transplant and/or have been re-transplanted.
  5. Patients taking immunosuppression for other diseases besides their liver transplant.
  6. Patients unable to give written informed consent in accordance with research ethics board guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Validation of Tolerance Gene Expression Profile | Enrollment to one year post cessation of immunosuppression
  The primary endpoint of this study is the identification and validation of a unique tolerance gene expression profile, consisting of a 6 gene profile, in 3-6 operationally tolerant patients compared to 25 rejecting and 25 healthy controls.

SECONDARY OUTCOMES:
Tolerance gene expression profile in graft versus peripheral blood mononuclear cells (PBMCs) | Enrollment to one year post cessation of immunosuppression
  This endpoint will be defined as the ratio of patients (n=55) that will express the tolerance gene expression profile in the liver graft versus in the peripheral blood mononuclear cells.
Test of tolerance gene expression profile | Enrollment to one year post cessation of immunosuppression
  This endpoint will assess whether the tolerance gene expression profile can be successfully used to select immunosuppressed patients for the successful weaning off immunosuppression. This endpoint will be evaluated using the number of successful immunosuppression-weaned patients from a 7-10 patient cohort. Successful immunosuppression-weaned patients are defined as patients who achieve an immunosuppression free state without any histological or clinical evidence of rejection for a minimum of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Levy, M.D., Principal Investigator — University Health Network, University of Toronto; Leslie Lilly, M.D., Study Chair — University Health Network, Toronto; Nazia Selzner, M.D. PhD., Study Chair — University Health Network, Toronto; Meaghan MacArthur, M.Ed, Study Director — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chruscinski A, Rojas-Luengas V, Moshkelgosha S, Issachar A, Luo J, Yowanto H, Lilly L, Smith R, Renner E, Zhang J, Epstein M, Grant D, McEvoy CM, Konvalinka A, Humar A, Adeyi O, Fischer S, Volmer FH, Taubert R, Jaeckel E, Juvet S, Selzner N, Levy GA. Evaluation of a gene expression biomarker to identify operationally tolerant liver transplant recipients: the LITMUS trial. Clin Exp Immunol. 2022 Jan 28;207(1):123-139. doi: 10.1093/cei/uxab011. PMID 35020854